CLINICAL TRIAL: NCT04693741
Title: Xenografts With Platelet-rich Fibrin Versus Autogenous Bone in Alveolar Cleft Grafting: A Comparative Clinical Study
Brief Title: Xenografts With Platelet-rich Fibrin Versus Autogenous Bone in Alveolar Cleft Grafting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hager Montaser Sayed Bedeer, MBBS, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: alveolar bone graft
Record Dates: First submitted 2020-10-27; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Alveolar Cleft

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two groups according to the surgical procedure performed as follows:
  Group A: the autogenous iliac bone graft will be used to fill the alveolar defect.
  Group B : Xenograft with PRF will be used to fill the alveolar defect.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autogenous iliac bone graft "group A" (Other): The autogenous iliac bone graft will be used to fill the alveolar defect.
  Interventions: Procedure: secondary alveolar bone graft; Procedure: Harvesting of the autogenous bone graft
- Xenograft with PRF "group B" (Other): Xenograft with PRF will be used to fill the alveolar defect.
  Interventions: Procedure: secondary alveolar bone graft; Procedure: Preparation of PRP

INTERVENTIONS:
Procedure: secondary alveolar bone graft — Under general anesthesia, the soft tissue in the gingiva surrounding the alveolar cleft will be injected with 0.5% lidocaine with 1:100,000 parts of epinephrine. At the alveolar cleft site, gingival sulcus incisions will be made on both sides of the cleft. The tissue will then elevated beneath the periosteum. The mucosa of the nasal floor and the oral mucosa will be dissected. Next, the bone particles will be implanted into the bone defect.
  Then, The cleft site will be closed without tension by the advancement of the gingival flaps.
Procedure: Harvesting of the autogenous bone graft — Under general anaesthesia ,the soft tissue in the superior iliac crest will injected with 0.5% lidocaine with 1:100,000 parts of epinephrine. The cancellous bone will harvested with an osteotome and then cut into small bone granules.
  Arms: Autogenous iliac bone graft "group A"
Procedure: Preparation of PRP — 10 ml of blood will be collected in vacuum tubes without anticoagulants which are then immediately centrifuged at a rate of 3000 rpm for 10 min. After centrifugation, the resultant product consists of three layers. The topmost layer consisting of acellular PPP (platelet poor plasma), PRF clot in the middle and RBCs at the bottom of the test tube. The attached red blood cells scraped off from it and discarded. The discarded PRF is then mixed with xenograft and placed inside the alveolar defect.
  Arms: Xenograft with PRF "group B"

SUMMARY:
this work aims to evaluate xenografts mixed with PRF versus autogenous bone graft in alveolar cleft grafting.

DETAILED DESCRIPTION:
The alveolar cleft is a maxillary bone defect resulting from incomplete fusion of the medial nasal process (MNP) and maxillary process (MXP) during embryonic development. Alveoloplasty may be classified as primary, secondary, and tertiary depending on the age of the patient. Literature defines primary when the alveoloplasty is performed at the same time as soft tissue repair. If performed at the age of 8 to 9 years before the eruption of the permanent canine, it is classified as secondary; it is classified as late secondary or tertiary if performed in the elderly. For patients with cleft lip and palate, secondary alveolar bone grafting (SABG) of the cleft alveolar ridge is performed when the patient has mixed dentition; SABG is a procedure that aims to create a bony bridge that restores dental arch continuity, repair the oronasal fistula, provide support to the structure of the alar base, facilitate subsequent orthodontic treatment, and promote tooth eruption. Autologous bone grafting is the gold standard for treating alveolar clefts, with the iliac crest bone being the most widely accepted donor site. Other materials such as growth factors, combinations of improved scaffolds and cell treatment/growth factors, biocomposites, and hemostatic agents can be used to regenerate bone and have been the subjects of intensive research.

ELIGIBILITY:
Inclusion Criteria:

* Age (7 - 12 years).
* Non-syndromic CLA or CLP.
* More than 6 months of follow-up.

Exclusion Criteria:

* History of previous alveolar surgery.
* History of active infection or underlying diseases such as hematologic disorders, neoplasm, and immune deficiency
* Patients who had received primary or tertiary ABG.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
measuring of bone volume 6 months post-operative. | 6 months
  Compare between outcome of xenografts mixed with PRF versus autogenous bone graft in alveolar cleft grafting regarding the newly formed bone volume.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Elshazly, professor, Principal Investigator — Assiut University; Awny asklany, doctor, Principal Investigator — Assiut University; mohammed nahed attia, doctor, Principal Investigator — Assiut University

REFERENCES:
- [Background] Moreau JL, Caccamese JF, Coletti DP, Sauk JJ, Fisher JP. Tissue engineering solutions for cleft palates. J Oral Maxillofac Surg. 2007 Dec;65(12):2503-11. doi: 10.1016/j.joms.2007.06.648. PMID 18022477
- [Background] Schnitt DE, Agir H, David DJ. From birth to maturity: a group of patients who have completed their protocol management. Part I. Unilateral cleft lip and palate. Plast Reconstr Surg. 2004 Mar;113(3):805-17. doi: 10.1097/01.prs.0000105332.57124.89. PMID 15108870
- [Background] Seifeldin SA. Is alveolar cleft reconstruction still controversial? (Review of literature). Saudi Dent J. 2016 Jan;28(1):3-11. doi: 10.1016/j.sdentj.2015.01.006. Epub 2015 Jun 25. PMID 26792963
- [Background] Seike T, Hashimoto I, Matsumoto K, Tanaka E, Nakanishi H. Early postoperative evaluation of secondary bone grafting into the alveolar cleft and its effects on subsequent orthodontic treatment. J Med Invest. 2012;59(1-2):152-65. doi: 10.2152/jmi.59.152. PMID 22450004
- [Background] Tan AE, Brogan WF, McComb HK, Henry PJ. Secondary alveolar bone grafting--five-year periodontal and radiographic evaluation in 100 consecutive cases. Cleft Palate Craniofac J. 1996 Nov;33(6):513-8. doi: 10.1597/1545-1569_1996_033_0513_sabgfy_2.3.co_2. PMID 8939379
- [Background] Kamal M, Ziyab AH, Bartella A, Mitchell D, Al-Asfour A, Holzle F, Kessler P, Lethaus B. Volumetric comparison of autogenous bone and tissue-engineered bone replacement materials in alveolar cleft repair: a systematic review and meta-analysis. Br J Oral Maxillofac Surg. 2018 Jul;56(6):453-462. doi: 10.1016/j.bjoms.2018.05.007. Epub 2018 May 30. PMID 29859781